CLINICAL TRIAL: NCT05209464
Title: A Mobile Tai Chi Platform for Fall Prevention and Cognition in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021P002665
Record Dates: First submitted 2022-01-08; First posted 2022-01-26 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Aging; Fall

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Tele-Tai Chi (Experimental): Study participants will follow a 12-week simplified Tele-Tai-Chi (TC) program delivered via a mobile application.
  Interventions: Device: Tele-Tai Chi

INTERVENTIONS:
Device: Tele-Tai Chi — Study participants will follow a 12-week simplified Tele-Tai-Chi (TC) program delivered via an application installed on a tablet. The intervention emphasizes essential TC movements that are easily comprehensible and can be performed repetitively in a flowing manner. The protocol includes up to six core TC movements based on the traditional Cheng Man-Ch'ing's Yang-style short form. Additionally, a set of traditional TC warm-up exercises that focus on loosening the physical body, incorporating mindfulness and imagery into movement, promoting overall relaxation, and coordinating breathing awareness are included. Chairs are used in the protocol for a subset of seated warm-up exercises, as well as for stability and rest as needed. Participants will be asked to practice the protocol (45-60 min) at home for at least 3 days a week for 12 weeks. The TC program will also include 2 or more live instructional sessions via Zoom with a TC instructor.

SUMMARY:
The investigators will assess feasibility and acceptability of the Tele-Tai Chi (TC) intervention; explore changes in clinically relevant outcome measures including: physical activity, self-efficacy, quality of life, cognitive function, balance, gait, and evaluate changes in TC proficiency. To achieve this, the investigators are running a single-arm study for older adults that involves a 12-week home-based Tai Chi intervention. Study participation includes four remote and/or in-person (at Spaulding Rehabilitation Hospital) visits to evaluate study participants (mobility tests and questionnaires).

DETAILED DESCRIPTION:
The overall goal of the study is to test the delivery of a novel Tele-Tai Chi (TC) intervention in a single-arm feasibility study for community-dwelling TC-naïve older adults. The investigators will assess feasibility and acceptability of the Tele-TC intervention and its specific components through both qualitative and quantitative feedback, as well as the systematic tracking of adherence data to inform future trials and potential clinical use of the Tele-TC system. The investigators will also explore changes in outcome measures including physical activity, self-efficacy, quality of life, cognition, balance and gait, and evaluate changes in TC proficiency.

Participants will be assessed at 4 timepoints over the course of the 12-week Tele-TC intervention: at baseline, at 4 weeks, at 8 weeks, and at 12 weeks.

Study participants will be instructed to train on their own at least three times a week and to participate in one-on-one live sessions with TC instructors two or more times during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 60 and 85 years old
* Naïve to Tai-Chi practice (never practiced TC)
* Montreal Cognitive Assessment (MoCA) score between 17 and 13.
* Self-reported ability to walk continuously for 15 minutes without an assistive device
* Working email address
* Prior experience with and current access to a computer, smart phone or tablet device

Exclusion Criteria:

* Chronic neuromuscular conditions (e.g. Parkinson's disease, multiple sclerosis, stroke)
* Acute medical conditions requiring hospitalization within the past 6 months or that could interfere with safely participating in the study
* Active cancer
* Significant musculoskeletal conditions requiring chronic use of pain medication
* Significant cognitive impairment (Diagnosed with dementia (self-reported), or Montreal Cognitive Assessment (MoCA)-Blind score < 13)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tele-Tai Chi
Started | 8
Completed | 7
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 70 [63 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Protocol Adherence
Description: The percentage of Tele-Tai-Chi practice sessions completed by participants.
Time Frame: Percentage at post-intervention (after 12 weeks)
Population: Data analysis was limited only to subjects who participated in the intervention and completed both baseline and post-intervention assessments.
Measure: Mean (Standard Deviation); unit: percentage of sessions completed
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
percentage of sessions completed | 78.6 (45.1)

2. Primary Outcome: Retention of Study Participants
Description: The percentage of participants who complete the study.
Time Frame: At study completion, 12 weeks from the beginning of the study
Population: Please note that 1 participant who was found not eligible after consent.
Measure: Number; unit: percentage of subjects retained
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 8
percentage of subjects retained | 87.5

3. Primary Outcome: System Usability Scale
Description: The scale is based on a 10-item questionnaire with five response options (from Strongly agree to Strongly disagree) in which participants rate the usability of the system. The scale ranges from 0 to 100, with higher scores indicating greater usability.
Time Frame: At post-intervention (after 12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
score on a scale | 87.9 (11.4)

4. Other Pre Specified Outcome: Ease of Use of the Tele-Tai Chi Platform (Qualitative Interview)
Description: Qualitative interview about ease of use of the Tele-Tai Chi platform.
Time Frame: At post-intervention (after 12 weeks)
Population: 1 of the 8 participants was found ineligible after providing consent. 1 additional participant did not provide feedback about the ease of use of the Tai Chi platform. The remaining 6 subjects provided positive feedback.
Measure: Number; unit: percentage of participants
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
percentage of participants | 100

5. Other Pre Specified Outcome: Activities-specific Balance Confidence (ABC) Scores
Description: This is 16-item self-report measure in which participants rate their balance confidence to perform motor activities. The minimum score is 0. The maximum score is 100. Positive changes (i.e., higher scores post-intervention) would represent a positive outcome.
Time Frame: Changes from baseline at 12 weeks (post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
score on a scale | 0.8 (11)

6. Other Pre Specified Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) 29 Scores
Description: The PROMIS 29 instrument is a 29-item questionnaire assessing each of the following domains: anxiety, depression, fatigue, physical function, pain interference, pain intensity, sleep disturbance, and ability to participate in social roles and activities. The minimum score is 4 per domain, except for pain intensity for which the minimum score is 0. The maximum score per domain is 20, except for pain intensity for which the maximum score is 10. For the physical function and the ability to participate in social roles and activities domains a high score is indicative of positive outcome. For the anxiety, depression, fatigue, sleep disturbance, pain interference, and pain intensity a low score is indicative of positive outcome.
Time Frame: Changes from baseline at 12 weeks (post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
score on a scale
  Ability to Participate in Social Roles/Activities | -0.7 (0.5)
  Anxiety/Fear | -0.7 (0.8)
  Depression/Sadness | -0.2 (1.3)
  Fatigue | -1.8 (1.9)
  Pain Interference | 0.7 (3.4)
  Physical Function | -0.2 (1.2)
  Sleep Disturbance | -1.2 (2.5)
  Pain Intensity | 0.2 (2.2)

7. Other Pre Specified Outcome: Physical Activity Scale for the Elderly (PASE)
Description: Self-reported level of physical activity in individuals aged 65 years or older during the previous 7 days. The score accounts for the type of activities performed and the time of performance of each activity. The minimum score is 0. The scale has theoretical maximum value of 864, if subjects spent 24 hours per day over 7 days engaged in vigorous activities. However, as this is not possible, a maximum value of 400 is typically considered as that would correspond to being engage in vigorous activities for 8 hours per day + more moderate activities for 4.5 hours per day.
Time Frame: Changes from baseline to post-intervention (at 12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
score on a scale | -10 (43.8)

8. Other Pre Specified Outcome: Trail Making Test A/B Scores
Description: The test to assess executive cognitive function. It has two parts: TMT A (number sequence only) considers visual search, and TMT B (alternating numbers and letters) evaluates executive control. The participant is asked to draw a line between 24 circles randomly arranged on a page that have to be linked in consecutive order. The TMT is scored by how long it takes to complete the test.
Time Frame: Changes from baseline at 12 weeks (post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
seconds
  Part A | -14.8 (22.6)
  Part B | -39 (44.4)

9. Other Pre Specified Outcome: Self-Efficacy Exercise (SEE) Questionnaire
Description: 9-item questionnaire that focuses on the self-efficacy expectations for exercise for older adults. The minimum score is 0. The maximum score is 90. Positive changes (i.e., higher scores post-intervention) would represent a positive outcome.
Time Frame: Changes from baseline at 12 weeks (post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
score on a scale | -2 (4.1)

10. Other Pre Specified Outcome: Change in Tai Chi Proficiency Score
Description: Tai Chi experts will use video recordings to score proficiency using a developed instrument to score each of the six Tai Chi movements performed by participants. The minimum score is 6. The maximum score is 30 per Tai Chi exercise. Positive changes (i.e., higher scores post-intervention) would represent a positive outcome. The change in Tai Chi proficiency score ranges from -24 to +24. A change equal to 0 represents no change in proficiency.
Time Frame: Changes from baseline at 12 weeks (post-intervention)
Population: 1 of the 8 participants was found ineligible after providing consent. 1 additional participant did not completed both baseline and post-intervention assessments. Data analysis was limited the remaining 6 participants completed both baseline and post-intervention assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
score on a scale | 6.1 (3.3)

11. Other Pre Specified Outcome: Timed-Up-and-Go
Description: Test routinely used in clinical practice to determine fall risk. The participant is asked to stand up from a chair, walk 3 meters, turns 180°, walk 3 meters back, and sits back down with back resting against the chair.
Time Frame: Changes from baseline at 12 weeks (post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 5
seconds | -1.69 (0.74)

12. Other Pre Specified Outcome: Timed-Up-and-Go Dual Task
Description: Test routinely used in clinical practice to determine fall risk and ambulation status. The participant is asked to stand up from a chair, walk 3 meters, turns 180°, walk 3 meters back, and sits back down with back resting against the chair while counting backwards by three.
Time Frame: Changes from baseline at 12 weeks (post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 5
seconds | -0.76 (6.45)

13. Other Pre Specified Outcome: Single Leg Stance
Description: Measured with a motion capture system. Balance on each leg (two trials): The participant is asked to stand on one leg for as long as they can up to a maximum of 30 seconds.
Time Frame: Changes from baseline at 12 weeks (post-intervention)
Population: Data analysis was limited only to subjects who participated in the intervention and completed both baseline and post-intervention assessments. Only the trial with the longest time was considered for analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
seconds
  Right Leg | 5.68 (4.43)
  Left Leg | 5.13 (11.5)

14. Other Pre Specified Outcome: Sit-to-Stand Performance
Description: Measure of fall risks. The participant is asked to stand up from a chair while keeping their arms crossed across their chest and repeat the task as many times as possible during a period of 30 seconds.
Time Frame: Changes from baseline at 12 weeks (post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: repetitions
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 5
repetitions | 1 (2)

15. Other Pre Specified Outcome: Postural Sway and Balance
Description: Participants are instructed to perform two tasks: 1) stand on both legs with feet shoulder-width apart for approximately 20 seconds, and 2) stand on both legs with feet close to each other again for approximately 20 seconds. A sensor positioned at the waist is used to track the displacement of the center of mass during the 20 second data collection (for each task). The root mean square (RMS) value of the acceleration data collected using the sensor positioned at the waist is estimated in the antero-posterior (AP) and medio-lateral (ML) directions for the middle 15 seconds of each experiment. Data is gathered at baseline and post-intervention and derived for each condition for a total of 8 variables.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: Data analysis was limited only to subjects who participated in the intervention and completed both baseline and post-intervention assessments. The root mean square (RMS) value of the acceleration in the antero-posterior (AP) and medio-lateral (ML) directions at the waist sensor was calculated for middle 15 seconds of each experiment (i.e., standing on both legs with feet shoulder-width apart and standing on both legs with feet close to each other).
Measure: Mean (Standard Deviation); unit: millimeters per second squared
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
millimeters per second squared
  Feet Apart AP - Baseline | 60 (0.7)
  Feet Apart AP - Post-Intervention | 60.4 (0.7)
  Feet Apart ML - Baseline | 60.4 (0.7)
  Feet Apart ML - Post-intervention | 60.4 (0.8)
  Feet Together AP - Baseline | 59.8 (0.6)
  Feet Together AP - Post-Intervention | 59.7 (0.5)
  Feet Together ML - Baseline | 59.7 (0.7)
  Feet Together ML - Post-intervention | 59.8 (0.6)

16. Other Pre Specified Outcome: Normalized-to-height Stride Length
Description: Study participants undergo an instrumented gait evaluation. Stride length is defined as the distance from ipsilateral foot contact to the next ipsilateral foot contact during gait. Normalized-to-height stride length is derived by computing the stride length and dividing such value by the height of the study participant.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
unitless
  Normalized Stride Length - Baseline (unitless) | 0.42 (0.02)
  Normalized Stride Length - Post-intervention (unitless) | 0.43 (0.04)

17. Other Pre Specified Outcome: Activity Level
Description: Physical activity (e.g. number of steps per day) derived using a wrist-worn activity monitor.
Time Frame: Changes from baseline at 12 weeks (post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
steps per day | 179 (2226)

18. Other Pre Specified Outcome: Mini-Balance Evaluation Systems Test (MiniBEST)
Description: MiniBEST Test: Test to assess dynamic balance. It is a 14-item test scored using a three-level ordinal scale. This test will be performed only in individuals who are willing to be tested in the laboratory (as opposed to via a remote visit). The minimum score is 0. The maximum score is 28. Positive changes (i.e., higher scores post-intervention) would represent a positive outcome.
Time Frame: Changes from baseline at 12 weeks (post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
score on a scale | -3 (3.1)

19. Other Pre Specified Outcome: Controlled Oral Word Association Test (COWAT) Scores
Description: The test examines working memory span. COWAT requires the participant to produce as many words as possible that begin with a given letter of the alphabet (F,A,S). There is 1 minute allowed for each of the three letters. The score is the sum of all acceptable words produced in the three trials.
Time Frame: Changes from baseline at 12 weeks (post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
words | 3 (2.2)

20. Other Pre Specified Outcome: Change in Digit Span Test Score
Description: The test assesses short-term memory by asking participants to memorize and recall in correct serial order a number of digits (i.e., numerals from 0 to 9). The test start asking participants to memorize fewer digits and then the number of digits is increased. The number sequences get progressively more difficult. Scores are based on the number of sequences correctly recalled (i.e., until the participant consecutively fails two trials of the same digit span length).
Time Frame: Changes from baseline at 12 weeks (post-intervention)
Population: Data analysis was limited only to subjects who participated in the intervention and completed both baseline and post-intervention assessments. Only the length of the longest sequence successfully completed was considered.
Measure: Mean (Standard Deviation); unit: sequences
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 5
sequences | 0.5 (0.58)

21. Other Pre Specified Outcome: Change in Grip Strength
Description: Investigators measure the grip strength of both upper limbs using a hand grip dynamometer. They repeat the measure three times (per side) for a total of six trials. The average value of the six trials is derived. Measures are gather at baseline and post-intervention. The difference in mean values (post-intervention minus baseline) is reported.
Time Frame: Changes from baseline at 12 weeks (post-intervention)
Population: Data analysis was limited only to subjects who participated in the intervention and completed both baseline and post-intervention assessments. The average of three trials was considered for the analysis.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
kilograms | 2.4 (2.1)

22. Other Pre Specified Outcome: Stride Time Variability
Description: Study participants undergo an instrumented gait evaluation. Stride time is measured as the time from foot contact to the next foot contact of the same leg. Stride time variability is defined as the standard deviation of the stride time values estimated for a session.
Time Frame: Baseline and post-intervention (approximately 12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Tele-Tai Chi
Number analyzed (Participants) | 6
milliseconds
  Stride Time Variability - Baseline | 7.86 (9.46)
  Stride Time Variability - Post-intervention | 3.83 (3.54)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the intervention period (approx. 12 weeks).
Arm/Group | Tele-Tai Chi
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tele-Tai Chi (N=7)
Delayed onset muscle pain (Musculoskeletal and connective tissue disorders) | 2 (2) — Several subjects reported muscle soreness. Some attributed the muscle soreness to physical activity, including practicing Tai Chi. All instances resolved without intervention.
Flu-like illness (Infections and infestations) | 2 (2) — Several subjects reported flu-like symptoms including sore throat and muscle soreness. All resolved without intervention.
Low back pain (Musculoskeletal and connective tissue disorders) | 2 (2) — Several subjects reported flares of pre-existing low back pain. None attributed the flares to the practice of Tai Chi. One was found to have a small, non-displaced fracture of the spine not requiring intervention. All symptoms returned to baseline.
Cholecystitis (Gastrointestinal disorders) | 1 (1) — One subject reported vague right-sided abdominal pain. Coincidentally, he was found to have an infection of the gallbladder during a hospitalization for flu-like symptoms. Was awaiting possible sugical resolution at study end.
Fall (Injury, poisoning and procedural complications) | 2 (2) — Several subjects reported falls, none were during the practice of Tai Chi. Falls did not result in hospitalization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT05209464/Prot_SAP_001.pdf